CLINICAL TRIAL: NCT06488963
Title: The Effect of Cold Therapy on Peripheral Neuropathy: A Pilot Randomized Controlled Trial
Brief Title: The Effect of Cold Therapy on Peripheral Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Eysan Hanzade Umac, research assistant, Koç University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KOCUNIVERSITY
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: The sample will consist of pediatric oncology patients aged 7 to 18 with select diagnoses (see inclusion criteria) who receive VCR. The G*Power software was used to analyze the sample's size (Faul et al., 2007). Since no similar previous study was identified, we aimed to reach a medium effect size for sample size calculation. Based on a medium effect size (f:0.40), 80% (1 - β error) power, and 95% (α error) confidence level within two groups and six repeated measurements, the sample size was calculated as 16 for each group, and a total of 32 children. Considering the expected dropout rate, the number was increased %10 and so 36 children will be recruited.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Children in the control group will receive standard care. VIPN is expected to follow at the end of the third cycle, nearly three months from the first VCR dose/application. Accordingly, no additional intervention will be performed to prevent peripheral neuropathy in children in the control group.
  Standard care: The clinic uses no pharmacological or non-pharmacological method as standard care for preventing VIPN. For patients with VIPN in the pediatric oncology clinic, dose reduction or treatment interruption is performed. Children will be excluded from the study if such a situation occurs during the research time period.
- Cold Therapy/Intervention Group (Experimental): In addition to standard care in the clinic, cold therapy will be applied to the children in the intervention group while they are receiving VCR in the inpatient pediatric oncology clinic. Children in the intervention group will wear cold therapy gloves and socks.To maintain the appropriate level of cold, the research assistant will replace the iced gel packs in the gloves and socks every 5 min during the treatment.
  Interventions: Other: NatraCure Cold Therapy gloves and socks

INTERVENTIONS:
Other: NatraCure Cold Therapy gloves and socks — These gloves and socks will be adjusted and tied to the child's wrists and ankles. There are sizes suitable for all ages and the dimensions of the gloves and socks can be adjusted with a snap fastener. The gloves and socks contain a soft Lycra lining and four inner gel cold packs to ensure full length cold therapy treatments. When the children wear these gloves and socks, they can still move their fingers and toes easily. In addition, it is a great advantage that the iced gel packs do not touch the child's skin directly.
  Arms: Cold Therapy/Intervention Group

SUMMARY:
This study examines the feasibility, acceptability, and efficacy of cold therapy on vincristine-induced peripheral neuropathy (VIPN) in pediatric patients with cancer.

Vincristine (VCR) is one of the most used vinca alkaloid chemotherapy in pediatric oncology patients. It leads to symptoms of peripheral neuropathy, numbness in the hands and feet, tingling, muscle/joint pain, burning sensation, decreased peripheral reflexes, and constipation. These symptoms negatively affect the daily life and quality of life of children. Therefore, it is essential to managing peripheral neuropathy. We aim to decrease the level of VIPN and pain and improve patients' quality of life.

Unfortunately, the neurotoxicity mechanisms of vinca alkaloids are not well known, which is one of the significant limitations in developing effective treatments to prevent VIPN among pediatric oncology patients. We were unable to locate a randomized controlled trial that has evaluated the effectiveness, tolerability, and acceptability of cold therapy on VIPN for pediatric oncology patients. Our study findings will be the first in Turkish national and international literature, and we believe that our results will provide evidence for clinical nursing practice.

DETAILED DESCRIPTION:
An estimated 400 000 children and adolescents ages 0-19 years old are diagnosed with cancer each year (WHO, 2021a). More than 80% of children with cancer are cured in high-income countries, where comprehensive care is generally available; whereas in some low- and middle-income countries less than 30% of patients survive (WHO, 2021b; Lam et al., 2019). Considering the global increase in childhood cancer incidence (Bhakta et al., 2019; Ward et al., 2019), it is critical to characterize the long-lasting side effects of treatment for childhood cancer and accurately assess, monitor, and ultimately develop management strategies to prevent treatment-related side effects (Kandula et al., 2016). Many chemotherapy agents used in cancer treatment can cause acute and chronic peripheral nervous system injury and dysfunction, termed chemotherapy-induced peripheral neuropathy (CIPN) (Rodwin et al., 2021; Kandula et al., 2016). CIPN is a significant problem becoming more prevalent as oncological therapies that use potentially neurotoxic chemotherapy enhance cancer cure and survival (Cavaletti et al., 2019). Peripheral neuropathy is a severe side effect of chemotherapeutic agents, and it can damage the sensory-motor-autonomic regions of the peripheral nervous system (Park et al., 2013; Kandula et al., 2016). Peripheral nerve toxicity has been described with vinca alkaloids, platinum compounds, taxanes, epothilones, bortezomib, and thalidomide (Kandula et al., 2016; Kandula et al., 2018; Cavaletti et al., 2019). Acute CIPN can develop during chemotherapy, necessitating dosage reduction or discontinuation and reducing survival (Colvin, 2019). In a recent systematic review of 42 publications (2009-2020) the reported CIPN incidence ranges from 2.8% to 100%, depending on risk variables. Sensory, motor, autonomic CIPN, and pain had incidence rates of 2-28%, 50-72%, 0.8-83%, and 5.7-44%, respectively (Smith et al., 2021). According to another review, although not life-threatening, CIPN threatens function in children and adolescents treated for cancer both during and following treatment (Bjornard et al., 2018). Smith et al. (2021) noted, "…sensory and motor neuropathy, pain, and functional impairments…" are not uncommon and appear to continue into adulthood. The most common CIPN symptoms in children and adolescents are numbness, tingling, neuropathic pain in the upper and lower limbs, weakness, loss of ankle dorsiflexion range of motion (foot drop), and impaired balance (van de Velde et al., 2017; Kandula et al., 2016; Schouten et al., 2020; van de Velde et al., 2021) VCR is one of the most commonly used vinca alkaloids in pediatric cancer patients and is included in a variety of multiple chemotherapy treatments for acute lymphoblastic leukemia, lymphomas, neuroblastoma, sarcomas, and central nervous system tumors (Mora et al., 2016; Schouten et al., 2020). Neurotoxicity as a prominent side effect of VCR, defined by autonomic and peripheral sensory-motor neuropathy, has been documented in three studies to be as low as 12% and as high as 87% of VCR-exposed children (Gilchrist et al., 2014; van de Velde et al., 2017; van de Velde et al., 2021). The fact that the prevalence of VIPN is so wide is due to the difference in the measurement tools used (van de Velde et al., 2017). VIPN symptoms generally arise after only a few VCR injections, and symptoms often fade a few months after VCR medication is stopped. Paresthesia, constipation, muscular weakness, areflexia, neuropathic pain, and lack of sensation symptoms commonly relate to VIPN (van de Velde et al., 2021).

VIPN treatment addresses symptoms and involves analgesics like gabapentin and amitriptyline (van de Velde et al., 2021). However, the only successful therapy option for VIPN is VCR dosage reduction, even though this limits optimal treatment (Mora et al., 2016). The limited treatment options for VIPN and the symptoms it causes in children have been linked to reducing the quality of life (QoL) both during and after treatment (Mora et al., 2016). Furthermore, it is known that peripheral neuropathy pain affects QoL during cancer therapy. However, it is uncertain how much VIPN affects the QoL in children with cancer during therapy (Bjornard et al., 2018; van de Velde et al., 2021).

Many pharmacological and non-pharmacological methods are used in the management of peripheral neuropathy. However, the neurotoxicity mechanisms of peripheral neuropathy are not well known, which a significant limitation in discovering effective treatments to prevent VIPN among pediatric oncology patients. A systematic review focusing on the efficacy and safety of cryotherapy for preventing VIPN in adults, reported that cryotherapy is a reasonable option to prevent VIPN (Bailey et al., 2021). The primary mechanism of benefit from cryotherapy has been hypothesized to be via vasoconstriction that decreases blood flow (and therefore, chemotherapy delivery) to treated areas (Loprinzi et al., 2020). Unfortunately, the following factors prevent the use of cryotherapy to prevent CIPN: (i) rare reports of frostbite, (ii) patient irritation, (iii) administrative difficulties (for patients, parents, and care professionals alike), and (iv) the lack of conclusive evidence that this approach reduces CIPN (Loprinzi et al., 2020). Nevertheless, many cryotherapy studies have shown the effectiveness of cryotherapy on peripheral neuropathy in adults (Beijers et al., 2020; Ng et al., 2020), we were unable to identify any studies in children and adolescents with cancer. There is a need for studies to evaluate the effectiveness of cryotherapy in reducing peripheral neuropathy in pediatric oncology patients. This study aims to evaluate the effectiveness, tolerability, and acceptability of cold therapy on VIPN among pediatric oncology patients in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* aged 7-18 years,
* receiving VCR therapy,
* diagnosed with leukemia, medulloblastoma, rhabdomyosarcoma, or Wilms tumor,
* able to speak and understand Turkish
* receiving initial treatment
* consent to participate in the research project.

Exclusion Criteria: Risk factors for peripheral neuropathy were considered exclusion criteria. Risk factor criteria were:

* receiving a dose of VCR <2.5 mg/m2,
* receiving VCR and azole antifungal treatment simultaneously,
* a hematological malignancy with neurological disease,
* a history of peripheral neuropathy,
* diabetes,
* self-reported cold sensitivity.
* Additionally, children who receive chemotherapy or other treatment using the peripheral veins of their hands or feet will not be included since the cold application is contraindicated.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
National Cancer Institute Common Terminology Criteria for Adverse Events v5 Peripheral Neuropathy Scale | Before starting each VCR application, the child's VIPN in the last week post the previous application will be evaluated. One week after the last VCR dose, the child's VIPN will be evaluated.
  The NCI CTCAE version 5.0 (ctep.cancer.gov) includes toxicity criteria for adverse events such as peripheral sensory and motor neuropathy, constipation, and neuralgia. The grading scale, used by health professionals is from 0-5, with 0=no toxicity and 5=death. In this study, a research assistant (PhD student in pediatric nursing) responsible for data collection will be trained to perform CTCAE scoring, review all medical records, and assign CTCAE version 5.0 sensory and motor scores according to the published criteria based on clinician documentation of signs and symptoms.

SECONDARY OUTCOMES:
Wong-Baker FACES® Pain Rating Scale | Before starting each VCR application, the child's pain in the last week post the previous application will be evaluated. One week after the last VCR dose, the child's pain will be evaluated.
  This scale consists of six facial expressions. Facial expressions range from 0 points "no pain-very happy" to 10 points "unbearable pain-crying" (Wong-Baker FACES Foundation, 2016). The self-report scale is commonly used for children aged 3-18 (Martin et al., 2018). It has good validity and reliability for measuring pain intensity (Ball et al., 2017), and is psychometrically appropriate and widely used in clinical practice (Stinson et al., 2006). The psychometric properties of this scale are also suitable for evaluation by parent proxy (Schiavenato, 2008). The scale has been translated into Turkish. (Wong-Baker FACES Foundation, 2016). For the present study, the Wong-Baker FACES® scale will be used for evaluating children's self-report and parental reports of the child's pain. This pain scale is commonly used in Turkey to evaluate children's pain. It is used as a standard measurement tool in the pain assessment of children aged 3-18 in all pediatric clinics in Turkey.

OTHER OUTCOMES:
Pediatric Quality of Life Inventory (PedsQL) 3.0 Cancer Module Survey | Before starting each VCR application, the child's QoL in the last week post the previous application will be evaluated. One week after the last VCR dose, the child's QoL will be evaluated.
  This scale was developed to measure the health-related QoL of children and adolescents aged 2-18 years (Varni et al., 2002). The reliability and validity of the Turkish Version of the PedsQL 3.0 Cancer Module testing was performed by Kabak et al. (2016). The PedsQL 3.0 Cancer Module was designed to measure pediatric cancer-specific health-related QoL. The 27-item multidimensional PedsQL 3.0 Cancer Module Acute Version encompasses 8 subscales: 1) pain and hurt (2 items), 2) nausea (5 items), 3) procedural anxiety (3 items), 4) treatment anxiety (3 items), 5) worry (3 items), 6) cognitive problems (5 items), 7) perceived physical appearance (3 items), and 8) communication (3 items). The child self-report and parent-proxy report are filled in considering QoL over the previous seven days.

CONTACTS AND LOCATIONS:
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No